CLINICAL TRIAL: NCT01861743
Title: Multimodal Analgesia Versus Routine Care Pain Management for Minimally Invasive Spine Surgery: A Prospective Randomized Study
Brief Title: Multimodal Analgesia Versus Routine Care Pain Management
Acronym: MMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: data was not collected accurately
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Frank M. Phillips, MD, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13020402
Record Dates: First submitted 2013-05-08; First posted 2013-05-24 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Degenerative Disc Disease Lumbar; Spinal Stenosis; Lumbar Spondylolisthesis
Keywords: Multi-modal Pain Management; Lumbar fusion; misTLIF
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multimodal analgesia (Experimental): multiple analgesic medications utilized in a synergistic manner to control pain while minimizing side-effects of individual drugs due to decreased doses. This includes pre-operative patient education, intra-operative pain management and post-operative pain protocols.
  Interventions: Other: Multimodal Analgesia
- Patient Controlled analgesia (Active Comparator): Pain management using patient controlled narcotic analgesia.
  Interventions: Other: Patient controlled analgesia

INTERVENTIONS:
Other: Multimodal Analgesia — Subjects are given medications preop, intraop and postop that implement a multi-modal approach to managing pain.
  Arms: Multimodal analgesia
Other: Patient controlled analgesia — Subjects will be treated with patient controlled narcotic analgesia for pain management.
  Arms: Patient Controlled analgesia

SUMMARY:
Most patients undergoing surgery experience significant post-operative pain. Inadequate peri-operative pain management may decrease post-operative mobilization and increase length of hospitalization. Additionally, poorly managed acute post-operative pain analgesia is associated with an increased risk of developing chronic pain and delayed wound healing.

Lumbar spine surgery is particularly painful, often requiring a multi-day hospitalization. The most common post-operative analgesia used in spine surgery is narcotic medication delivered via an intravenous patient controlled analgesia (IV PCA).

A multimodal peri-operative pain management protocol for spine surgery has the potential to not only decrease pain but also to improve recovery, decrease narcotic consumption, decrease length of stay in the hospital and reduce both direct and indirect hospital costs.

The purpose of this study is to determine if post-operative pain and rate of recovery are improved in patients undergoing spine surgery using MMA compared to usual analgesic care.

DETAILED DESCRIPTION:
We hypothesize patients undergoing spinal fusion who receive peri-operative MMA will have:

1. decreased post-operative pain compared to patients receiving usual care for pain management.
2. shorter hospital LOS compared to patients receiving usual care pain management.
3. fewer analgesic-related post-operative complications (urinary retention, ileus, etc) compared to patients receiving usual care pain management.
4. improved physical functioning at the time of hospital discharge compared to patients receiving usual care pain management.
5. better short and long term outcomes. Subjects will be randomized to MMA (Group 1) or usual care (Group 2). The unit of randomization will be a week (Monday through Sunday). Each week will randomly be assigned to MMA or usual care. Subjects who are hospitalized into a consecutive week will continue with the pain regimen they were assigned upon hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing single level MIS-TLIF
* Patients able to provide informed consent

Exclusion Criteria:

* Allergies or other contraindications to medicines in the protocol
* Current liver disease with documented liver function test abnormality
* Current renal disese with documented glomerular filtration rate (GFR) < 60 mL/min/1.73m2
* Baseline (pre-operative) opioid use greater than 30 mg of morphine equivalents/day
* Active alcohol dependence
* Active illicit drug dependence

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2016-12-31 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Numeric pain scale | Patients will be followed post-operatively while in the hospital (Avg 1-3 days), and a 6 weeks, 3 months, 6 months, 1 year and 2 years.
  (a) While in the hospital, patients' pain is assessed by a nurse-driven protocol. Assessments are every four to six hours, within 60 minutes after receiving an intravenous pain medication and within 90 minutes of receiving an oral pain medication. This assessment includes rating subjective rating of ones pain on a verbal numeric rating scale (NRS) of 0-10. The maximum pain score for each post-operative day will be compared.

SECONDARY OUTCOMES:
Patient satisfaction | Post operatively (avg: 1-3 days)
  At each pain assessment (minimum every 4 hours), partients are asked if they are satisfied with their pain management. (yes/no)

OTHER OUTCOMES:
Length of Stay | Post operatively (avg: 1-3 days)
Discharge destination | Post operatively (avg:1-3 days)
  Determine whether patients are discharged to home or to another facility (e.g. rehab, etc)
Adverse events | Post operatively (avg: 1-3 days)
Disease specific and General health outcome measures | Pre operatively (within 1 month of date of surgery) and Post operatively (6 weeks, 3months, 6 months, 1 year and 2 years)
  Short form 36 and the Oswestry Disabilty Index

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Phillips, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center-Orthopedic Spine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kim JC, Choi YS, Kim KN, Shim JK, Lee JY, Kwak YL. Effective dose of peri-operative oral pregabalin as an adjunct to multimodal analgesic regimen in lumbar spinal fusion surgery. Spine (Phila Pa 1976). 2011 Mar 15;36(6):428-33. doi: 10.1097/BRS.0b013e3181d26708. PMID 21372654
- [Result] Rajpal S, Gordon DB, Pellino TA, Strayer AL, Brost D, Trost GR, Zdeblick TA, Resnick DK. Comparison of perioperative oral multimodal analgesia versus IV PCA for spine surgery. J Spinal Disord Tech. 2010 Apr;23(2):139-45. doi: 10.1097/BSD.0b013e3181cf07ee. PMID 20375829